CLINICAL TRIAL: NCT02950168
Title: Edoxaban Management in Diagnostic and Therapeutic Procedures
Acronym: EMIT-AF/VTE
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DSE-EDO-02-15-EU
Record Dates: First submitted 2016-10-28; First posted 2016-10-31 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Atrial Fibrillation; Venous Thromboembolism
Keywords: Diagnostic procedures; Interventional procedures; Planned or unplanned; Edoxaban-treated population
MeSH Terms: conditions — Atrial Fibrillation; Venous Thromboembolism | interventions — edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Edoxaban: All patients treated with edoxaban with a planned or unplanned diagnostic or interventional procedure
  Interventions: Procedure: Edoxaban

INTERVENTIONS:
Procedure: Edoxaban — Edoxaban according to Summary of Product Characteristic (SMPC)
  Other Names: Lixiana

SUMMARY:
Patients receiving Novel Oral Anticoagulation (NOACs) undergo diagnostic and therapeutic procedures at a rate of 10% per year. Short half-lives and rapid onset of action allow for short periods of NOAC interruption without heparin bridging. There is only minimal information on the peri-procedural usage pattern of edoxaban and the related outcome data currently available. Therefore, further real-world clinical data on the peri-procedural usage pattern of edoxaban within any diagnostic or interventional procedure in patients with non-valvular atrial fibrillation (NVAF) or venous thromboembolism (VTE) will be collected in this registry.

DETAILED DESCRIPTION:
Patients treated with edoxaban and with a planned or unplanned diagnostic or interventional procedure will be enrolled in this study in order to evaluate the peri-procedural dosing of edoxaban in patients with diagnostic or therapeutic procedures and collect details of the type diagnostic or therapeutic procedures. Patients from 7 different countries and care settings (primary care, secondary care, and different medical specialties) will be enrolled. The study will last until approximately 2000 procedures have been documented, e.g., until about 2000 participants are enrolled, which is expected to take approximately 2.5 years. Any relevant diagnostic or interventional procedure reported will be collected and documented in the electronic case report form (eCRF). Patients will be followed for 30 days after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients taking edoxaban for a therapeutic indication for edoxaban according to SMPC including NVAF, DVT or PE
* Patients with a planned or unplanned diagnostic or therapeutic procedure
* Written informed consent
* Availability of patients for follow-up by telephone by the site
* No concurrent participation in an interventional study (simultaneous participation in other non-interventional studies is possible)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Edoxaban-treated patients with NVAF, VAT or PE undergoing planned or unplanned diagnostic or interventional procedures
Sampling Method: Non-Probability Sample
Enrollment: 1197 (Actual)
Dates: Start 2016-11; Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with major bleeding within 30 days after a planned or unplanned procedure | within 30 days after a procedure
Percentage of participants with clinically-significant non-major bleeding (CRNMB) within 30 days after a planned or unplanned procedure | within 30 days after a procedure
  Categories: minor bleeding, all bleeding, and death from any cause

SECONDARY OUTCOMES:
Percentage of participants with acute coronary syndromes within 30 days after a planned or unplanned procedure | within 30 days after a procedure
  Categories: unstable angina pectoris, myocardial infarction, non-haemorrhagic stroke, transient ischaemic attack (TIA), systemic embolism (SEE), deep vein thrombosis (DVT), pulmonary embolism (PE) and cardiovascular (CV) mortality

OTHER OUTCOMES:
Number of procedures undergone by trial participants by type | within the 2.5 year study
  Categories: Planned and Unplanned

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Background] Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, Waldo AL, Ezekowitz MD, Weitz JI, Spinar J, Ruzyllo W, Ruda M, Koretsune Y, Betcher J, Shi M, Grip LT, Patel SP, Patel I, Hanyok JJ, Mercuri M, Antman EM; ENGAGE AF-TIMI 48 Investigators. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2013 Nov 28;369(22):2093-104. doi: 10.1056/NEJMoa1310907. Epub 2013 Nov 19. PMID 24251359
- [Result] Vranckx P, Valgimigli M, Eckardt L, Tijssen J, Lewalter T, Gargiulo G, Batushkin V, Campo G, Lysak Z, Vakaliuk I, Milewski K, Laeis P, Reimitz PE, Smolnik R, Zierhut W, Goette A. Edoxaban-based versus vitamin K antagonist-based antithrombotic regimen after successful coronary stenting in patients with atrial fibrillation (ENTRUST-AF PCI): a randomised, open-label, phase 3b trial. Lancet. 2019 Oct 12;394(10206):1335-1343. doi: 10.1016/S0140-6736(19)31872-0. Epub 2019 Sep 3. PMID 31492505
- [Derived] Unverdorben M, Colonna P, Jin J, Kohler S, Santamaria A, Saxena M, Borrow A, Chen C, von Heymann C, Vanassche T. Periprocedural Edoxaban Management and Clinical Outcomes in Patients Undergoing Transcatheter Cardiovascular Procedures in the EMIT-AF/VTE Program. Clin Appl Thromb Hemost. 2024 Jan-Dec;30:10760296241260728. doi: 10.1177/10760296241260728. PMID 38881370
- [Derived] von Heymann C, Unverdorben M, Colonna P, Santamaria A, Saxena M, Vanassche T, Kohler S, Borrow AP, Jin J, Chen C. Management of edoxaban therapy and clinical outcomes in patients undergoing major or nonmajor surgery: a subanalysis of the EMIT-AF/VTE study. Thromb J. 2023 Dec 14;21(1):124. doi: 10.1186/s12959-023-00568-2. PMID 38098072
- [Derived] Santamaria A, Chen C, Colonna P, von Heymann C, Saxena M, Vanassche T, Jin J, Unverdorben M. Predictive Factors and Clinical Events Associated with Edoxaban Interruption and Heparin Bridging Strategy: EMIT-AF/VTE. Clin Appl Thromb Hemost. 2023 Jan-Dec;29:10760296231200223. doi: 10.1177/10760296231200223. PMID 37697813
- [Derived] Unverdorben M, von Heymann C, Santamaria A, Saxena M, Vanassche T, Jin J, Laeis P, Wilkins R, Chen C, Colonna P. Elderly patients with atrial fibrillation in routine clinical practice-peri-procedural management of edoxaban oral anticoagulation therapy is associated with a low risk of bleeding and thromboembolic complications: a subset analysis of the prospective, observational, multinational EMIT-AF study. BMC Cardiovasc Disord. 2020 Dec 1;20(1):504. doi: 10.1186/s12872-020-01766-w. PMID 33256590